CLINICAL TRIAL: NCT00723983
Title: A Phase I, Open Label, Single-Dose, Four-Way Crossover Study Comparing the Pharmacokinetics of NP101 (Sumatriptan Iontophoretic Transdermal Patch) With an Oral Formulation of Imitrex® (50mg) in Migraine Subjects During an Acute Migraine Attack and During a Non-Migraine Period
Brief Title: Phase I, Open Label, Single-Dose, Four Way Crossover Study to Compare the PK of NP101 With Oral Imitrex® (50mg) in Migraine Subjects During an Acute Migraine Attack and During a Non-Migraine Period
Acronym: NP101-011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuPathe Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PROT-15-NP101-011
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Period 1 (Active Comparator): Subject dosed with oral sumatriptan succinate during an acute migraine attack.
  Interventions: Drug: Sumatriptan succinate
- Period 2 (Active Comparator): Subject dosed with oral sumatriptan during a non-migraine period.
  Interventions: Drug: Sumatriptan succinate
- Period 3 and Period 6 (Experimental): Subject dosed with NP101 during an acute migraine attack.
  Interventions: Drug: NP101 Study Patch
- Period 4 and Period 5 (Experimental): Subject dosed with NP101 study patch during a non-migraine period.
  Interventions: Drug: NP101 Study Patch

INTERVENTIONS:
Drug: Sumatriptan succinate — Sumatriptan succinate 50 mg taken orally
  Arms: Period 1; Period 2
Drug: NP101 Study Patch — NP101 study patch 4 hour application
  Arms: Period 3 and Period 6; Period 4 and Period 5

SUMMARY:
To compare the pharmacokinetics of NP101 with a currently approved oral formulation of Imitrex® (50 mg) in migraine subjects both during an acute migraine attack and during a non-migraine period.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects, between the ages of 18 to 65 years.
* Subjects with a diagnosis of migraine headache, with or without aura, as defined in the ICHD-II, and the diagnosis was made before the age of 50.
* The majority of a subject's headaches during a migraine attack are moderate to severe in intensity.
* Subject has history of regularly occuring migraines, accompanied by nausea or vomiting.
* Subject has at least one year history of migraine based upon subject testimony.
* Subject will be judged to be in good health, based upon the results of a medical history, physical examination, vital signs, ECG and laboratory profile.
* Subjects must voluntarily sign and date and Informed Consent agreement approved by an IRB.
* Subject must have a negative drug screen and re-screen.
* Female subjects of childbearing potential must have a negative pregnancy test at Screening and Re-Screening.
* Subject has two acceptable patch application sites.

Exclusion Criteria:

* Subject has or plans to start stop, or change treatment (including dose change) of any medication within one month prior to the subject screening date and through the end of study.
* Subject has less than 2 migraines per month or subject has more than 15 headache days/month for any of the 3 months prior ot screening.
* Subject who has suspected or confirmed cardiovascular disease that contraindicates study participation.
* Subject has history of epilepsy or conditions associated with lower seizure threshold.
* Subject with Raynaud's disease.
* Subject with hemiplegic or basilar migraine.
* Subject with a current diagnosis of major depressive disorder.
* Subject who has taken non-triptan serotonergic drugs including SSRI's, SNRI, TCAs or MAOI's or preparations containing St. John's Wort within month prior to screening and/or is planning to start any of these medications during the study and through the End of Study Visit.
* Subject is unwilling to discontinue use of PD5 inhibitors (eg. Viagra, Levitra, Cialis) from screening through End of Study Visit.
* Subject with a history of significant allergy or hypersensitivity to any component of the NP101 study patch.
* Subject who has any generalized skin irritation or disease including eczema, psoriasis, melanoma, acne or contact dermatitis.
* Subject has a positive test result for hepatitis B, hepatitis C or is known to be HIV positive.
* Subjects with moderate or severe hepatic dysfunction defined as SGOT/AST or SGPT/ALT ≥ 2 times the upper limit of normal range, or alkaline phosphatase or total bilirubin ≥ 1.5 times the upper limit of normal range or if in the opinion of the investigator, the subject's history, physical examination or other laboratory tests suggest hepatic dysfunction.
* Female subjects who are pregnant, breast feeding, or if not of childbearing potential, is not using or is unwilling to use an effective form of contraception during the study and for a period of 30 days following final dosing.
* Subjects with a known history of tolerability issues with sumatriptan.
* Subject who is considered by the investigator or NuPathe to be an unsuitable candidate for this study.
* Subject has a history (within 1 year) or current evidence of drug or alcohol abuse or dependence.
* Subject has participated in a clinical study within 30 days of Screening or is planning to participate in another clinical study.
* Subject has clinically significant abnormal labs, vital signs or ECG
* Subject is electrically sensitive or who has an implantable electronic device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Compare the pharmacokinetics of NP101 with a currently approved formulation of Imitrex in migraine subjects during an acute migraine attack and during a non-migraine period. | PK samples at pre and 0.25, 0.5, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 10, 12 and 24 hours post each dose/period for Periods 1, 2, 3, and 4 [24 hour PK will not be done for Periods 5 and 6]

CONTACTS AND LOCATIONS:
Overall Officials: Kerri L Wilks, MD, CPI, Principal Investigator — MD clinic
Locations (1):
- MD Clinic, Hallandale, Florida, United States